CLINICAL TRIAL: NCT02303158
Title: Study of the Relationship Between Protein Biomarkers in Cerebrospinal Fluid and the Risk of Progression to Alzheimer&Apos;s Disease in a Cohort of Patients With Depression
Brief Title: Relationship Between Protein Biomarkers in Cerebrospinal Fluid and Alzheimer&Apos;s Disease in Patients With Depression
Acronym: LIDEAL
Status: Terminated | Type: Observational
Why Stopped: futility of the sample
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Other Study IDs: IISPV-LIDEAL-HTVC
Record Dates: First submitted 2014-05-30; First posted 2014-11-27 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Biomarkers; Depression; dementia; cerebrospinal fluid; neuropsychological
MeSH Terms: conditions — Alzheimer Disease; Depression; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid (CSF), blood serum, blood plasma and whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is currently accepted that depression during midlife is a risk factor for Alzheimer's disease (AD). Furthermore, several prospective population studies have demonstrated that depression is an independent risk factor for incident dementia of different types (e.g. vascular, mixed, Alzheimer's disease). However, it is not clear, what are the mechanisms that link depression and dementia, and if depression can be a prodromal manifestation of AD. There are also studies that suggest that depression could be an initial sign of AD.

Objective:

1. Demonstrate that late life depression (over 60 years of age) constitutes the first manifestation of AD.
2. Define by rating scales and life stressors have differential risk profiles evolutionary AD.
3. To study the relationship between the subtypes of depression and CSF biomarkers, neurophycological test and evolution to AD.

DETAILED DESCRIPTION:
Groups of subjects: patients with recent apparition of late life depression without fulfilling the dementia criteria (Global Deterioration Scale, GDS, stages 1, 2 and 3). A longitudinal, prospective population study with two years follow-up. A cohort of will be included in the study. The patient's depression will be defined and categorized according to its severity (Yesavage Scale), whether it's endogenous or reactive (Holmes and Rahe scale) and taking into account the patient's medical history of depression.

There will be a prospective follow-up of conversion to dementia (starting from GDS Stage 4). It will be considered that dementia corresponds to AD if the biological markers of LCR present typical changes of AD at the moment of inclusion (Beta amyloid low and P-tau high).

It will be studied if there's any correlation between the clinically defined depression types and a high risk of progression to dementia and especially to AD.

ELIGIBILITY:
Inclusion Criteria:

* >= 60 years.
* GDS (Reisberg Gobal Dementia Scale) of 2 to 3.
* Geriatric Depression Scale of Yesavage >=12.
* History of previous depressive episodes resolved, but the emotional situation 15 months before inclusion, necessarily have to be normal.

Exclusion Criteria:

* Established dementia of any cause, or secondary degenerative dementia of any origin
* Primary diagnosis of cognitive impairment with psychiatric illness (schizophrenia , bipolar disorder, personality disorders ... )
* Dual diagnosis of chronic depression, dysthymia more than 15 months duration, or major depression with psychotic or atypical symptoms
* Neuroimaging with significant chronic vascular involvement
* To take drugs with known side effects on cognition and it is suspected that the neuropsychological deficits.
* Moderate or severe sensory deprivation or functional illiteracy in the neuropsychological study can not be performed
* Neoplastic diseasesContraindication to performing a lumbar puncture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive patients referred from Primary Care and Psychiatry, Neurology with consultations for specialist for cognitive impairment and / or depression who met the inclusion criteria of the study assessment.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Analysis of cerebrospinal fluid | between the second and the fifth day after inclusion visit
  Measure alterations in amyloid AB 1-42, total tau protein and phosphorylated tau protein, in pg/ml. Those alterations will be correlated with the evolution to dementia at final visit (after 24 months +/- 5 days)

SECONDARY OUTCOMES:
Conversion to dementia | first measure at inclusion visit and second measure at final visit (after 24 months +- 5 days).
  Measure increases scores in Global Dementia Scale (GDS), considering no dementia GDS from 1 until 3, and evolution to dementia GDS form 3 until 6
Depression subtypes | at basal visit
  classify the type of depression by scores in two scales. One of them is Yesavage with scores between 11-17 corresponding with "low depression" and scores between 18-30 with "major depression". the second ones is Vital Stressors Scale of Holmes and Rahe which define adaptative depression as scores upper than 150 and non adaptative depression as scores between 0 and 150.
  Subtype of depression will be correlated with posterior evolution to dementia at final visit (after 24 months +/- 5 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Tortosa, Verge de la Cinta, Tortosa, Tarragona, Spain

REFERENCES:
- [Result] Tam CW, Lam LC. Association between late-onset depression and incident dementia in Chinese older persons. East Asian Arch Psychiatry. 2013 Dec;23(4):154-9. PMID 24374487
- [Result] Gracia-Garcia P, de-la-Camara C, Santabarbara J, Lopez-Anton R, Quintanilla MA, Ventura T, Marcos G, Campayo A, Saz P, Lyketsos C, Lobo A. Depression and incident Alzheimer disease: the impact of disease severity. Am J Geriatr Psychiatry. 2015 Feb;23(2):119-29. doi: 10.1016/j.jagp.2013.02.011. Epub 2013 Jun 20. PMID 23791538
- [Result] Diniz BS, Butters MA, Albert SM, Dew MA, Reynolds CF 3rd. Late-life depression and risk of vascular dementia and Alzheimer's disease: systematic review and meta-analysis of community-based cohort studies. Br J Psychiatry. 2013 May;202(5):329-35. doi: 10.1192/bjp.bp.112.118307. PMID 23637108
- [Result] Wallin K, Bostrom G, Kivipelto M, Gustafson Y. Risk factors for incident dementia in the very old. Int Psychogeriatr. 2013 Jul;25(7):1135-43. doi: 10.1017/S1041610213000409. Epub 2013 Apr 11. PMID 23574921
- [Result] Rosenberg PB, Mielke MM, Appleby BS, Oh ES, Geda YE, Lyketsos CG. The association of neuropsychiatric symptoms in MCI with incident dementia and Alzheimer disease. Am J Geriatr Psychiatry. 2013 Jul;21(7):685-95. doi: 10.1016/j.jagp.2013.01.006. Epub 2013 Feb 6. PMID 23567400
- [Result] Nozaki S, Yoshimura K, Mimura M. [Depression and dementia: perspectives from clinical studies]. Brain Nerve. 2012 Dec;64(12):1387-97. Japanese. PMID 23209065
- [Result] Potter GG, Wagner HR, Burke JR, Plassman BL, Welsh-Bohmer KA, Steffens DC. Neuropsychological predictors of dementia in late-life major depressive disorder. Am J Geriatr Psychiatry. 2013 Mar;21(3):297-306. doi: 10.1016/j.jagp.2012.12.009. PMID 23395197
- [Result] Gao Y, Huang C, Zhao K, Ma L, Qiu X, Zhang L, Xiu Y, Chen L, Lu W, Huang C, Tang Y, Xiao Q. Depression as a risk factor for dementia and mild cognitive impairment: a meta-analysis of longitudinal studies. Int J Geriatr Psychiatry. 2013 May;28(5):441-9. doi: 10.1002/gps.3845. Epub 2012 Jul 19. PMID 22815126 (Retraction: PMID 25914914 Int J Geriatr Psychiatry. 2015 Apr;30(4):435)
- [Result] Dubois B, Feldman HH, Jacova C, Hampel H, Molinuevo JL, Blennow K, DeKosky ST, Gauthier S, Selkoe D, Bateman R, Cappa S, Crutch S, Engelborghs S, Frisoni GB, Fox NC, Galasko D, Habert MO, Jicha GA, Nordberg A, Pasquier F, Rabinovici G, Robert P, Rowe C, Salloway S, Sarazin M, Epelbaum S, de Souza LC, Vellas B, Visser PJ, Schneider L, Stern Y, Scheltens P, Cummings JL. Advancing research diagnostic criteria for Alzheimer's disease: the IWG-2 criteria. Lancet Neurol. 2014 Jun;13(6):614-29. doi: 10.1016/S1474-4422(14)70090-0. PMID 24849862